CLINICAL TRIAL: NCT06155019
Title: Switch From Etravirine to Doravirine as a Part of Antiretroviral Combination in Virologically Suppressed People Living With HIV (PLWH): the French Multicenter, Observational SWEED Study
Brief Title: Switch From Etravirine to Doravirine as a Part of Antiretroviral Combination
Acronym: SWEED
Status: Completed | Type: Observational
Sponsor: Centre de Recherches et d'Etude sur la Pathologie Tropicale et le Sida (Other)
Responsible Party: Sponsor
Other Study IDs: CREPATS 16
Record Dates: First submitted 2023-11-24; First posted 2023-12-04 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non comparative: switch from etravirine to doravirine, with no change in associated antiretroviral drugs, will be assessed retrospectively

SUMMARY:
The main objective of the SWEED study is to determine whether doravirine containing ART is able to maintain viral suppression at W48 in HIV-1 infected people living with HIV (PLWH) receiving etravirine containing ART:

* An ARV strategy containing doravirine as a replacement for etravirine can maintain virological suppression in participants with controlled viral replication under ARV treatment containing etravirine, with a virological success rate >90%
* This strategy can maintain virological suppression even in the event of NNRTI resistance mutations acquired in the past
* This strategy is well tolerated
* The emergence of resistance to NNRTIs is uncommon in the event of virological failure under the ARV regimen containing doravirine

DETAILED DESCRIPTION:
The evolution of HIV infection from fatal to chronic has been enabled by advances in development and access of antiretroviral treatment (ART), which has also resulted in life expectancy of PLWH approaching that of those uninfected.In addition, over the past few years, new drugs and news regimens have offered improved efficacy, safety and tolerability. The 95-95-95 UNAIDS target, i.e. to diagnose 95% of PLWHIV (1st 95), provide ART to 95% of those diagnosed with HIV (2nd 95), and to reach viral suppression in 95% of patients on ART (3rd 95), is being achieved in several countries. Calls to add a fourth target, i.e. to improve the quality of life for PLWHIV, have grown stronger since the concept was introduced in 2016. The twin aims are long-term treatment durability and improved quality of life with a focus on personalized treatment.

Switching or simplifying ART in the setting of HIV suppression may improve pill burden, dosing frequency, safety, tolerability, and/or food requirements. At times, ART switch or simplification is elective, such as consolidating a multiple-tablet to a single-tablet regimen (STR). Other times, it is necessary to eliminate drug-drug interactions (DDIs) and/or minimize active or potential treatment-associated adverse events (AEs). The fundamental principle of switching or simplifying ART is to preserve virologic suppression without jeopardizing future ART options.

Etravirine, a second generation NNRTI, has been demonstrated to be effective on HIV strains with prior resistance mutations on reverse transcriptase impacting other NNRTIs, such as nevirapine, efavirenz or rilpivirine. It has even been used in salvage therapy, in association with darunavir and raltegravir, in uncontrolled patients with multiresistant strains. Etravirine is mostly prescribed twice daily, and is a strong enzymatic inducer providing many DDIs, complicating its use.

Doravirine, a last generation NNRTI, is approved in treatment-naïve and experienced HIV-infected individuals. In the DRIVE-FORWARD study, doravirine 100 mg QD, in combination with either TDF/FTC or ABC/3TC, achieved high virologic success at week 48 and was non-inferior to DRV/r + 2 NRTIs regardless of baseline HIV-RNA. In the DRIVE-AHEAD study, in treatment-naïve adults with HIV-1 infection, doravirine + 3TC/TDF administered once daily demonstrated a high antiviral potency with non-inferior efficacy to EFV/FTC/TDF regardless of baseline HIV-RNA, and a low rate of resistance, with only 1.6% of participants developing resistance to any study drug through W48. For virologically suppressed patients considering a change in therapy, switching to DOR/3TC/TDF was shown to be a well-tolerated option which was non-inferior to continuation of the previous regimen, with high rates of virologic suppression and low rates of virologic rebound. Long term results from the DRIVE-SHIFT trial showed that doravirine maintained virologic suppression and was generally well tolerated through 144 weeks of treatment. DOR/3TC/TDF as switch therapy showed a favorable lipid profile compared with previous regimens and results in minimal weight gain. The convenience achieved through switching to a DOR based regimen serves to achieve regimen simplification and could respond to patient demands for increased tolerability.

The DOR resistance profile is distinct from that of other NNRTIs with the in vitro selection of mutations at reverse transcriptase (RT) positions 106, 108, 188, 227, 230, 234 and 236. In vitro studies have also suggested that DOR has activity against viruses with certain mutations selected by other NNRTIs, including the K103N and Y181C mutations. In the DRIVE-SHIFT trial, conducted in virologically suppressed patients, 24 participants had a virus with baseline NNRTI mutations (K103N, Y181C and G190A) and 23/24 who switched to DOR/3TC/TDF remained virologically suppressed at the 48-week follow-up. This suggests that the most frequent NNRTI mutations at RT mutation positions 103, 181 and 190 probably not impact DOR activity in vivo.

Due to its virological properties, we believe that doravirine can advantageously replace etravirine, maintaining control of viral replication, in combination with other antiretrovirals, in virologically controlled patients, despite possible exposure to NNRTIs in the pass. Furthermore, doravirine is taken as a single tablet once a day, and causes almost no drug interactions, unlike etravirine.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* With HIV-1 infection
* On a regimen containing etravirine QD or BID combined with at least one other antiretroviral from any class except NNRTI
* Who had switched for a regimen containing doravirine combined with the same number of other antiretrovirals
* With plasma HIV-RNA <50 copies/mL for at least 12 months (one blip <200 copies/mL permitted) at time of switch to doravirine
* With at least 2 available pVL after the switch, and at least 48 weeks between the switch and the last available pVL*
* Who gave their non-opposition for the study

  * For patients who stopped doravirine-based treatment or were lost to follow-up before 48 weeks, only the theoretical duration of follow-up will be taken into account (time between the switch and the date of analysis)

Exclusion Criteria:

- Subject under " sauvegarde de justice " (judicial protection due to temporarily and slightly diminished mental or physical faculties), or under legal guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This observational, non-interventional, multicenter study will assess the efficacy of switching etravirine to doravirine in virally suppressed PLWH on stable etravirine containing ART, with at least 48 weeks of follow-up
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2023-12-08 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Measure the virological efficacy at week 48 a doravirine-containing ART to assess the effectiveness of the switch to maintain the virological success to W48 | 12 months
  Measure of plasma viral load assessed by RNA quantification using COBAS 6800 system (Roche)

CONTACTS AND LOCATIONS:
Overall Officials: Romain PALICH, DR, Principal Investigator — Pitie-Salpetriere Hospital, Infectious Diseases department
Locations (1):
- Pitié-Sapêtrière Hospital, Paris, France